CLINICAL TRIAL: NCT04566744
Title: NeuroCognitive Bases of Tool Use
Acronym: TECHNITION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Université Lumière Lyon 2 (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0677; 2020-A02115-34 (Other: ID-RCB)
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Tool use; fMRI; neuroimaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical tool use, tool making and construction (Experimental): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when solving mechanical problems in using either a physical tool, making a physical tool or building a construction. Only the fMRI experimental session is necessary. These experimental conditions related to the BOLD measures given by the fMRI technique will allow us to draw hypotheses on the neurocognitive mechanisms at work when we use or make physical tools as well as when we build constructions.
  Interventions: Other: fRMI
- Use of modern physical tools and stone tools (Experimental): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when solving mechanical problems in using either a modern physical tool or a stone tool. Only the fMRI experimental session is necessary. These experimental conditions related to the BOLD measures given by the fMRI technique will allow us to draw hypotheses on the neurocognitive mechanisms at work when we use or make physical tools irrespective of whether they are modern or old (i.e., stone tools).
  Interventions: Other: fRMI
- Use of modern physical, arbitrary and digital tools (Experimental): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when watching video clips of individuals using either a modern physical tool, an arbitrary tool (e.g., a washing machine) or a digital tool (e.g., a touchscreen). Only the fMRI experimental session is necessary. These experimental conditions related to the BOLD measures given by the fMRI technique will allow us to draw hypotheses on the neurocognitive mechanisms at work when we observe others using different kinds of tools, which have appeared progressively over technological evolution.
  Interventions: Other: fRMI
- Physical tool use and Internet (Experimental): The fMRI experimental conditions in this arm will allow us to study the activity of the brain when estimating the capacity to solve a mechanical problem with modern physical tools either alone or with the help of a Internet Tutorial. Only the fMRI experimental session is necessary. These experimental conditions related to the BOLD measures given by the fMRI technique will allow us to draw hypotheses on the neurocognitive mechanisms at work when we imagine and estimate solving a mechanical problem alone or with the help of the Internet;
  Interventions: Other: fRMI

INTERVENTIONS:
Other: fRMI — The measurements performed will be the participant's brain activity, as well as behavioral measurements associated with the tasks performed (response time, correctness of the response). Brain activity measurements will be performed on the Siemens 3T system of the MRI department of CERMEP. The subject will perform the task under study while the level of brain activity is recorded. The functional examination will be subdivided into several parts according to its total length in order to spare the subject. The total duration of MRI acquisitions will be approximately 1 hour regardless of the axis.

SUMMARY:
Tool use is considered to be the hallmark of complex cognitive adaptations that humans have achieved trough evolution, that provides an adaptive advantage to the human species. Even if nonhuman species do use tools too, human tool use is much more complex and sophisticated. If humans have special abilities for tool use, it has to be grounded in a specific neuroanatomical substrate. Humans and nonhumans share a similar prehension system located within the superior parietal lobe and the intraparietal sulcus. However, there is a human specificity: the supramarginal gyrus within the left inferior parietal lobe is unique to humans, and could play a central role in tool use. This project aims to study the neurocognitive bases of human tool use with functional Magnetic Resonance Imaging (fMRI), to precise the cognitive mechanisms through which humans are able to use tools.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18 and 65 years old
* Having given an informed consent for the study

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Persons under curators or deprived of civil rights or deprived of their freedom
* Not being registered with the French Social Security System
* Not able to read/write the French
* Neurologic or psychiatric illness, known or revealed during the inclusion visit
* Substance intake ( taking psychoactive medications or recreational drugs) on the day of the experiment
* Noise intolerance
* Unable to fill a questionnaire (severe cognitive troubles)
* Not willing that their personal doctor to be informed in case of a MRI anomaly.
* Not willing to be informed in case of MRI anomaly
* Subjects must not have metallic or electronic implants in the body : pacemakers or pacemaker wires, open heart surgery, artificial heart valve, brain aneurysm surgery, middle ear implant, hearing aid, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, or artificial limb or joint o foreign metallic objects in the body (bullets, pellets, shrapnel, or metalwork fragments) or current or past employment as machinists, welders or metal workers, tattoos near the head or neck regions, permanent makeup
* Not willing to complete the study
* Appearance of a exclusion criterion during the protocol
* Appearance of an undesirable event preventing the completion of the protocol
* Too great head movements (>4mm for the session)
* Detection of artifacts in the brain images collected

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygenation Level Dependent measure | 1 hour
  The primary outcome measure will be the Blood Oxygenation Level Dependent measure (BOLD) as permitted with functional Magnetic Resonance Imaging.This BOLD level will be collected for every voxel in the imaged brain, and at regular time intervals (TR = 3s) during the experimental session (about one hour). This is standard procedure for fMRI experiments. FMRI measures brain activity by detecting changes associated with blood flow. This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases. The primary form of fMRI uses the BOLD contrast in response to an experimental condition (Ogawa, Lee, Kay, & Tank, 1990), allowing researchers to track changes in oxygen consumption on the brain and therefore brain activity. BOLD effefct is computed by assessing the different relaxation times (T1 and T2) in the brain, as T1 and T2 are different in function of regional cerebral blood flows

CONTACTS AND LOCATIONS:
Overall Officials: François OSIURAK, PhD, Principal Investigator — Université Lyon 2
Locations (1):
- CERMEP, Bron, France